CLINICAL TRIAL: NCT05931042
Title: Neoadjuvant Therapy With Trastuzumab and Chemotherapy and the Resultant Pathologic Complete Response Observed in HER2 Positive Breast Cancer;a Systematic Review
Status: Completed | Type: Observational
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Maham Leeza Adil, Dr Maham Leeza Adil, Rawalpindi Medical College
Other Study IDs: 823678
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: HER2+ Breast Cancer
MeSH Terms: interventions — Trastuzumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group recieving Trastuzumab + Chemotherapy: Two different treatment regimens of Trastuzumab were giving in the 9 studies Dosage of trastuzumab was 4 mg/kg loading dose followed by 2 mg/kg every 3 weeks in four clinical trials included in this systematic review Dosage of trastuzumab was 8 mg/kg loading dose, followed by 6 mg/kg every 3 weeks in five clinical trials included in this systematic review The different chemotherapeutic agents given included Paclitaxel, docetaxel, fluorouracil, epirubicin, carboplatin, cyclophosphamide, methotrexate, and fluorouracil.
  Interventions: Drug: Trastuzumab
- Group receiving chemotherapy: Different neoadjuvant chemotherapy regimens were given in the nine clinical trials included in this systematic review. The different chemotherapeutic agents given included Paclitaxel, docetaxel, fluorouracil, epirubicin, carboplatin, cyclophosphamide, methotrexate, and fluorouracil.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab was given at dosage of either 4mg/kg or 8mg/kg at mostly a weekly interval (but differs among the different studies)

SUMMARY:
The goal of this systematic review is to assess the effectiveness of neoadjuvant chemotherapy and Trastuzumab in achieving pathological complete response (pCR) in patients with HER2-positive breast cancer. The main questions it aims to answer are:

* What is the overall rate of pathological complete response (pCR) in HER2-positive breast cancer patients treated with neoadjuvant chemotherapy and Trastuzumab?
* Are there any variations in the definition of pCR among the included trials?

Participants in the selected clinical trials were HER2-positive breast cancer patients with non-metastatic operable, locally advanced, or inflammatory breast cancer. The main tasks participants were asked to do and the treatments they received are as follows:

* Undergo neoadjuvant chemotherapy: Participants received chemotherapy treatment before their primary surgery.
* Receive Trastuzumab: Participants were administered Trastuzumab, a targeted therapy for HER2-positive breast cancer.

Researchers would compare the group of participants receiving neoadjuvant chemotherapy and Trastuzumab to other groups, if present, to see if there are differences in the rates of pathological complete response (pCR) or other effects.

DETAILED DESCRIPTION:
This systematic review aimed to assess the effectiveness of neoadjuvant chemotherapy and Trastuzumab in achieving pathological complete response (pCR) in patients with HER2-positive breast cancer. The researchers identified nine clinical trials that met the inclusion criteria. These trials included patients with non-metastatic operable, locally advanced, or inflammatory breast cancer, and they evaluated the pCR as the primary or secondary endpoint.

The trials utilized different chemotherapy and targeted therapy regimens, along with varying dosages of Trastuzumab. The primary outcome of interest was the pCR rate, while other survival outcomes were not analyzed. Among the 1,209 patients who received neoadjuvant chemotherapy and Trastuzumab, the overall pCR rate was found to be 42%.

The review provided detailed information about the design of the selected trials, patient characteristics, disease staging, HER2 status, administered treatment regimens, and primary/secondary endpoints. It also mentioned slight variations in the definition of pCR across the trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer that was found to be HER2 positive were included
* Only patients who underwent neoadjuvant therapy were included
* All cytotoxic chemotherapy regimens were considered eligible for this systematic review given that the same drugs were given at the same dose in every trial.

Exclusion Criteria:

* Patients with metastatic breast cancer were not included in the systematic review
* Results from adjuvant therapy were excluded from this study.
* Only the most recent publication (and the most informative) was included if numerous publications of the same trial were retrieved or if there was a case mix between publications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients found to have HER2+ breast cancer were included
Study Population: This study only included clinical trials. The review methods were decided before the start of the review. Studies that used the pathological complete response (pCR) as their primary or secondary endpoint were considered. The proportion of patients without invasive breast and axillary cancer was the criteria used to define pCR (ypT0/is and ypN0).
  Patients with breast cancer that was found to be HER2 positive were included. If the HER2 FISH test score was 2 or higher or the immunohistochemistry score for HER2 was +3, the HER2 status was interpreted as positive.
Sampling Method: Probability Sample
Enrollment: 1209 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 5 years
  5 trials labelled pCR as the absence of residual invasive cancer in the breast and lymph nodes while 4 trials defined pCR as the absence of invasive neoplastic cells at microscopic examination of the primary tumour at surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rawalpindi Medical University, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
No patient data to be shared

REFERENCES:
- [Background] I-SPY2 Trial Consortium; Yee D, DeMichele AM, Yau C, Isaacs C, Symmans WF, Albain KS, Chen YY, Krings G, Wei S, Harada S, Datnow B, Fadare O, Klein M, Pambuccian S, Chen B, Adamson K, Sams S, Mhawech-Fauceglia P, Magliocco A, Feldman M, Rendi M, Sattar H, Zeck J, Ocal IT, Tawfik O, LeBeau LG, Sahoo S, Vinh T, Chien AJ, Forero-Torres A, Stringer-Reasor E, Wallace AM, Pusztai L, Boughey JC, Ellis ED, Elias AD, Lu J, Lang JE, Han HS, Clark AS, Nanda R, Northfelt DW, Khan QJ, Viscusi RK, Euhus DM, Edmiston KK, Chui SY, Kemmer K, Park JW, Liu MC, Olopade O, Leyland-Jones B, Tripathy D, Moulder SL, Rugo HS, Schwab R, Lo S, Helsten T, Beckwith H, Haugen P, Hylton NM, Van't Veer LJ, Perlmutter J, Melisko ME, Wilson A, Peterson G, Asare AL, Buxton MB, Paoloni M, Clennell JL, Hirst GL, Singhrao R, Steeg K, Matthews JB, Asare SM, Sanil A, Berry SM, Esserman LJ, Berry DA. Association of Event-Free and Distant Recurrence-Free Survival With Individual-Level Pathologic Complete Response in Neoadjuvant Treatment of Stages 2 and 3 Breast Cancer: Three-Year Follow-up Analysis for the I-SPY2 Adaptively Randomized Clinical Trial. JAMA Oncol. 2020 Sep 1;6(9):1355-1362. doi: 10.1001/jamaoncol.2020.2535. PMID 32701140
- [Background] Ismael G, Hegg R, Muehlbauer S, Heinzmann D, Lum B, Kim SB, Pienkowski T, Lichinitser M, Semiglazov V, Melichar B, Jackisch C. Subcutaneous versus intravenous administration of (neo)adjuvant trastuzumab in patients with HER2-positive, clinical stage I-III breast cancer (HannaH study): a phase 3, open-label, multicentre, randomised trial. Lancet Oncol. 2012 Sep;13(9):869-78. doi: 10.1016/S1470-2045(12)70329-7. Epub 2012 Aug 9. PMID 22884505
- [Background] Buzdar AU, Ibrahim NK, Francis D, Booser DJ, Thomas ES, Theriault RL, Pusztai L, Green MC, Arun BK, Giordano SH, Cristofanilli M, Frye DK, Smith TL, Hunt KK, Singletary SE, Sahin AA, Ewer MS, Buchholz TA, Berry D, Hortobagyi GN. Significantly higher pathologic complete remission rate after neoadjuvant therapy with trastuzumab, paclitaxel, and epirubicin chemotherapy: results of a randomized trial in human epidermal growth factor receptor 2-positive operable breast cancer. J Clin Oncol. 2005 Jun 1;23(16):3676-85. doi: 10.1200/JCO.2005.07.032. Epub 2005 Feb 28. PMID 15738535
- [Background] Buzdar AU, Suman VJ, Meric-Bernstam F, Leitch AM, Ellis MJ, Boughey JC, Unzeitig G, Royce M, McCall LM, Ewer MS, Hunt KK; American College of Surgeons Oncology Group investigators. Fluorouracil, epirubicin, and cyclophosphamide (FEC-75) followed by paclitaxel plus trastuzumab versus paclitaxel plus trastuzumab followed by FEC-75 plus trastuzumab as neoadjuvant treatment for patients with HER2-positive breast cancer (Z1041): a randomised, controlled, phase 3 trial. Lancet Oncol. 2013 Dec;14(13):1317-25. doi: 10.1016/S1470-2045(13)70502-3. Epub 2013 Nov 13. PMID 24239210
- [Background] Semiglazov V, Eiermann W, Zambetti M, Manikhas A, Bozhok A, Lluch A, Tjulandin S, Sabadell MD, Caballero A, Valagussa P, Baselga J, Gianni L. Surgery following neoadjuvant therapy in patients with HER2-positive locally advanced or inflammatory breast cancer participating in the NeOAdjuvant Herceptin (NOAH) study. Eur J Surg Oncol. 2011 Oct;37(10):856-63. doi: 10.1016/j.ejso.2011.07.003. Epub 2011 Aug 16. PMID 21843921
- [Background] van Ramshorst MS, van Werkhoven E, Mandjes IAM, Schot M, Wesseling J, Vrancken Peeters MTFD, Meerum Terwogt JM, Bos MEM, Oosterkamp HM, Rodenhuis S, Linn SC, Sonke GS. Trastuzumab in combination with weekly paclitaxel and carboplatin as neo-adjuvant treatment for HER2-positive breast cancer: The TRAIN-study. Eur J Cancer. 2017 Mar;74:47-54. doi: 10.1016/j.ejca.2016.12.023. Epub 2017 Feb 10. PMID 28335887
- [Background] Gianni L, Pienkowski T, Im YH, Roman L, Tseng LM, Liu MC, Lluch A, Staroslawska E, de la Haba-Rodriguez J, Im SA, Pedrini JL, Poirier B, Morandi P, Semiglazov V, Srimuninnimit V, Bianchi G, Szado T, Ratnayake J, Ross G, Valagussa P. Efficacy and safety of neoadjuvant pertuzumab and trastuzumab in women with locally advanced, inflammatory, or early HER2-positive breast cancer (NeoSphere): a randomised multicentre, open-label, phase 2 trial. Lancet Oncol. 2012 Jan;13(1):25-32. doi: 10.1016/S1470-2045(11)70336-9. Epub 2011 Dec 6. PMID 22153890
- [Background] Shao Z, Pang D, Yang H, Li W, Wang S, Cui S, Liao N, Wang Y, Wang C, Chang YC, Wang H, Kang SY, Seo JH, Shen K, Laohawiriyakamol S, Jiang Z, Li J, Zhou J, Althaus B, Mao Y, Eng-Wong J. Efficacy, Safety, and Tolerability of Pertuzumab, Trastuzumab, and Docetaxel for Patients With Early or Locally Advanced ERBB2-Positive Breast Cancer in Asia: The PEONY Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Mar 1;6(3):e193692. doi: 10.1001/jamaoncol.2019.3692. Epub 2020 Mar 12. PMID 31647503
- [Background] Beitsch P, Whitworth P, Baron P, Rotkis MC, Mislowsky AM, Richards PD, Murray MK, Pellicane JV, Dul CL, Nash CH, Stork-Sloots L, de Snoo F, Untch S, Lee LA. Pertuzumab/Trastuzumab/CT Versus Trastuzumab/CT Therapy for HER2+ Breast Cancer: Results from the Prospective Neoadjuvant Breast Registry Symphony Trial (NBRST). Ann Surg Oncol. 2017 Sep;24(9):2539-2546. doi: 10.1245/s10434-017-5863-x. Epub 2017 Apr 26. PMID 28447218